CLINICAL TRIAL: NCT06715150
Title: NON-SURGICAL TREATMENT of PERI-IMPLANTITIS with or WITHOUT SYSTEMIC AZITHROMYCIN: a RANDOMIZED CLINICAL TRIAL in HUMANS
Brief Title: Non-Surgical Treatment of Peri-implantitis with Systemic Azithromycin or Placebo
Acronym: NSTP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Juan Blanco Carrión, Associate Professor, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USC77/2024; Self founding (Other: Universidade de Santiago de Compostela)
Record Dates: First submitted 2024-11-11; First posted 2024-12-04 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Peri-implantitis
Keywords: Non-surgical treatment; Azithromycin; Systemic antibiotic
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azithromycin 500 mg (Active Comparator): Systemic antibiotic: Azithromycin 500 mg every 24 hours for 3 days
  Interventions: Drug: Azithromcyin
- Placebo (Placebo Comparator): Same shape, size and dosage as test
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Azithromcyin — Immediately after the end of non surgical treatment of periimplantitis and depending on the result of randomization, the exact number of tablets of the placebo to be taken during the following days will be given to the patient.
  Arms: Azithromycin 500 mg
Other: Placebo — Immediately after the end of non surgical treatment of periimplantitis and depending on the result of randomization, the exact number of tablets of the placebo to be taken during the following days will be given to the patient.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the change in probing depth in patients with peri-implantitis, assessing the influence of systemic antibiotic (azithromycin) adjunctive to non-surgical treatment at 12 months. The secondary objective is to assess clinical, radiographic, microbiological, and systemic changes at 3, 6, and 12 months.

This study is designed as a placebo-controlled, randomized, triple-blind clinical trial in subjects diagnosed with peri-implantitis.

The treatment will consist of debridement of the implant surface and curettage of the pocket epithelium. The control group will receive placebo (1 placebo tablet per day for 3 days), and the test group will receive systemic azithromycin 500 mg per day for 3 days (1 tablet of 500 mg azithromycin per day for 3 days).

DETAILED DESCRIPTION:
Peri-implantitis is defined as the pathological alteration associated with plaque that occurs in the tissues surrounding dental implants, characterized by inflammation of the peri-implant mucosa and subsequent progressive loss of supporting bone. Bacterial colonization of the implant surface in a susceptible subject is considered the primary etiological factor of this pathology. Case series and clinical trials have demonstrated an additional benefit when using systemic antibiotics such as ornidazole or metronidazole after non-surgical treatment of peri-implantitis.

The rationale for conducting this clinical trial lies in the lack of randomized studies that have tested the non-surgical treatment of peri-implantitis with shorter antibiotic regimens and their potential impact on systemic health.

The primary objective of this randomized clinical trial is to evaluate the change in probing depth at 12 months in patients with peri-implantitis, assessing the influence of systemic antibiotic (azithromycin) as an adjunct to the non-surgical treatment of peri-implantitis.

The secondary objective is to assess clinical, radiographic, and microbiological changes at 3, 6, and 12 months. Additionally, systemic biomarkers, complete blood count, glycosylated hemoglobin and creatinine will be evaluated at day 7, and 3, 6, and 12 months. Endothelial function (endothelium-dependent vasodilation measured in the brachial artery) and subclinical atherosclerosis (measurement of carotid artery intima-media thickness) will be evaluated at 12 months.

Design: This research is designed as a 1-year randomized controlled trial (RCT), with 2 parallel groups, triple-blind, and placebo-controlled.

Population: Patients who come to the Periodontology Department, Faculty of Dentistry, University of Santiago de Compostela with dental implants presenting pathology.

Treatment Groups: Study group: patients treated by non-surgical treatment in conjunction with systemic azithromycin. Control group: patients treated by non-surgical treatment in conjunction with a placebo. Subjects will be randomly assigned to one of the two treatment groups.

Randomization: A balanced randomization by blocks will be performed to avoid imbalances between the two treatment groups. The randomization outcome will be stored in envelopes along with the antibiotic or placebo containers that will be delivered on the day of the non-surgical treatment.

Treatment: After the diagnosis of peri-implantitis, patients were instructed in oral hygiene and motivation was reinforced. After that, one session of nonsurgical treatment consisting of supra- and submucosal mechanical debridement using ultrasound with a metal periodontal tip was performed with concomitant irrigation of chlorhexidine of 0.12%. The tip removed granulation tissue and also touched the implant surface. After that, a steel curette Columbia 4R/4L was used to remove granulation tissue and minor mucosa curettage. If oral hygiene was not allowed by prosthetic design, a contour correction was made. Immediately after treatment, patients were prescribed to apply a chlorhexidine gel in the area 2 times a day for 2 weeks and depending on the result of randomization, the exact number of antibiotic or placebo tablets to be taken by the patient in the following days will be provided.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years;
* absence of systemic pathology contraindicating treatment;
* presence of at least 1 implant diagnosed with peri-implantitis: presence of bleeding on probing, probing depth ≥6 mm, and radiographic bone level ≥3 mm apical to the most coronal portion of the intraosseous part of the implant;
* absence of implant mobility;
* patients without periodontitis or with treated periodontitis;
* patients who understand the treatment and are willing to comply with it by providing written informed consent.

Exclusion Criteria:

* smokers ≥10 cigarettes/day;
* diabetic patients (HbA1c level ≥6,5%);
* pregnant or breastfeeding women;
* use of antibiotics, corticosteroids, and/or immunosuppressive treatment in the 3 months prior to the start of the study;
* allergy to azithromycin;
* patients with a history of bisphosphonate treatment;
* chronic consumption of non-steroidal anti-inflammatory drugs;
* bone loss exceeding the apex of the implant;
* prosthesis that does not allow access to peri-implantitis treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2026-01-10 (Estimated); Study Completion 2027-01-10 (Estimated)

PRIMARY OUTCOMES:
Change in probing depth | From enrollment to the end of treatment at 12 months
  The change in probing depth (quantitative dependent variable) at 12 months will be measured in millimeters as the distance from the mucosal margin to the bottom of the peri-implant pocket, using a millimetric CP15 UNC Hu-Friedy probe. The change in probing depth will also be measured at 3 and 6 months.

SECONDARY OUTCOMES:
Recession | From enrollment to the end of treatment at 12 months
  Distance from the implant shoulder to the margin of the peri-implant mucosa, measured in millimeters using a millimetric CP15 UNC Hu-Friedy probe. If the margin of the peri-implant mucosa is located apically to the implant shoulder, it will be recorded as a positive value (+); conversely, if the margin of the peri-implant mucosa is located coronally to the implant shoulder, it will be recorded as a negative value (-)
Clinical attachment level | From enrollment to the end of treatment at 12 months
  Distance from the implant shoulder to the bottom of the peri-implant pocket (probing depth + recession) measured in millimeters using a millimetric CP15 UNC Hu-Friedy probe
Bleeding index | From enrollment to the end of treatment at 12 months
  0: absent bleeding / 1: present bleeding
Plaque index | From enrollment to the end of treatment at 12 months
  0: absent plaque / 1: present plaque
Width of the keratinized mucosa | From enrollment to the end of treatment at 12 months
  From the peri-implant mucosal margin to the mucogingival line measured in millimeters using a millimetric CP15 UNC Hu-Friedy probe
Changes in radiographic bone level | From enrollment to the end of treatment at 12 months
  Distance from the implant shoulder to the apical extent of the bone defect in mesial, distal, and total (calculated as the average of mesial and distal distances) of each implant on standardized periapical radiographs following the long cone paralleling technique with individualized positioning devices.
Change in bacterial load | From enrollment to the end of treatment at 12 months
  The levels of the following pathogens will be determined: Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythia, Treponema denticola, Prevotella intermedia, Parvimonas micra, Fusobacterium nucleatum, Campylobacter rectus, Eikenella corrodens, Candida albicans and the total bacterial count.
Implant survival | From enrollment to the end of treatment at 12 months
  Maintenance of each implant's function included in the study
Endothelial function | From enrollment to the end of treatment at 12 months
  Measured by endothelium-dependent vasodilation in the brachial artery using a vascular ultrasound
Subclinical atherosclerosis | From enrollment to the end of treatment at 12 months
  Measured by the intima-media thickness of the carotid artery using a vascular ultrasound
Concentration of inflammatory cytokines biomarkers | From enrollment to the end of treatment at 12 months
  The predetermined biomarkers to be analyzed include a multiplex inflammatory panel (IL-1β, IL-12p70, IFN-γ, IL-6, IL-10, IL-8, TNF-α), measured in pg/mL
Concentration of endothelial activation/injury markers | From enrollment to the end of treatment at 12 months
  Endothelial activation/injury markers (E-selectin, P-selectin, thrombomodulin, ICAM-1, ICAM-3, VCAM-1), measured in ng/mL
Concentration of serum C-reactive protein | From enrollment to the end of treatment at 12 months
  C-reactive protein (CRP), measured in mg/L using Meso Scale assays (pro-inflammatory 7-PLEX, Vascular Injury Panel I, and V-PLEX Panel II)
Concentration of serum amyloid A | From enrollment to the end of treatment at 12 months
  Serum amyloid A (SAA), measured in µg/mL using Meso Scale assays (pro-inflammatory 7-PLEX, Vascular Injury Panel I, and V-PLEX Panel II)
Concentration of circulating blood cells | From enrollment to the end of treatment at 12 months
  Circulating blood cells will be measured in 10³/µL
Concentration of high-sensitivity CRP | From enrollment to the end of treatment at 12 months
  High-sensitivity CRP (hs-CRP) will be assessed using ELISA, in mg/L
Rate of lipid fractions | From enrollment to the end of treatment at 12 months
  Lipid fractions (triglycerides, total cholesterol, HDL, LDL) will be assessed in mg/dL using standard biochemical methods
Treatment success | From enrollment to the end of treatment at 12 months
  Treatment success will be established as achieving a probing depth ≤5 mm, without bleeding in more than one point, and without suppuration, in each implant included in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Blanco Carrión, Principal Investigator — Universidade de Santiago de Compostela
Locations (1):
- Department of Surgery and Medical-Surgical Specialties, Teaching and Research Unit in Periodontology. Faculty of Medicine and Dentistry, University of Santiago de Compostela., Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Orlandi M, Pranno N, Patel V, Papi P, Di Murro B, Pompa G, Polimeni A, Letizia C, Suvan J, D'Aiuto F. Peri-implant diseases and systemic inflammation: A preliminary analysis from a cross-sectional survey of patients with hypertension. J Periodontol. 2024 Jun;95(6):525-534. doi: 10.1002/JPER.21-0338. Epub 2024 May 14. PMID 38742572
- [Background] Blanco C, Linares A, Dopico J, Pico A, Sobrino T, Leira Y, Blanco J. Peri-implantitis, systemic inflammation, and dyslipidemia: a cross-sectional biochemical study. J Periodontal Implant Sci. 2021 Oct;51(5):342-351. doi: 10.5051/jpis.2100920046. PMID 34713995
- [Background] Linares A, Pico A, Blanco C, Blanco J. Adjunctive Systemic Metronidazole to Nonsurgical Therapy of Peri-implantitis with Intrabony Defects: A Retrospective Case Series Study. Int J Oral Maxillofac Implants. 2019 Sep/Oct;34(5):1237-1245. doi: 10.11607/jomi.7343. PMID 31528867
- [Background] Renvert S, Lessem J, Dahlen G, Renvert H, Lindahl C. Mechanical and repeated antimicrobial therapy using a local drug delivery system in the treatment of peri-implantitis: a randomized clinical trial. J Periodontol. 2008 May;79(5):836-44. doi: 10.1902/jop.2008.070347. PMID 18454662
- [Background] Linares A, Sanz-Sanchez I, Dopico J, Molina A, Blanco J, Montero E. Efficacy of adjunctive measures in the non-surgical treatment of peri-implantitis: A systematic review. J Clin Periodontol. 2023 Jun;50 Suppl 26:224-243. doi: 10.1111/jcpe.13821. Epub 2023 May 4. PMID 37143407
- [Background] Estefania-Fresco R, Garcia-de-la-Fuente AM, Egana-Fernandez-Valderrama A, Bravo M, Aguirre-Zorzano LA. One-year results of a nonsurgical treatment protocol for peri-implantitis. A retrospective case series. Clin Oral Implants Res. 2019 Jul;30(7):702-712. doi: 10.1111/clr.13456. Epub 2019 Jun 1. PMID 31090974
- [Background] Blanco C, Pico A, Dopico J, Gandara P, Blanco J, Linares A. Adjunctive benefits of systemic metronidazole on non-surgical treatment of peri-implantitis. A randomized placebo-controlled clinical trial. J Clin Periodontol. 2022 Jan;49(1):15-27. doi: 10.1111/jcpe.13564. Epub 2021 Oct 28. PMID 34713471